CLINICAL TRIAL: NCT00669799
Title: Topical Antibiotic Use In Chronic Rhinosinusitis A Double-Blinded, Randomized, Placebo Controlled Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: UNABLE TO PROCEED WITH STUDY DUE TO STAFFING OF COLLABORATIVE INVESTIGATORS
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Lockey, Principal Investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEIGS
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): clyndamyacin
  Interventions: Drug: gentamyacin
- 2 (Experimental): gentamicin
  Interventions: Drug: gentamyacin

INTERVENTIONS:
Drug: gentamyacin — topical internasal
  Arms: 1
Drug: gentamyacin — intranasal
  Arms: 2

SUMMARY:
Chronic rhinosinusitis is a pervasive and costly disease. Recent estimates describe over 20 million Americans suffering from this diagnosis at a cost of over $4.3 billion per year. Primary intervention consists of oral antibiotics and nasal steroid sprays. A role for antifungal irrigation has also been proposed. Topical antibiotics are used by some physicians, but there are few reports in the published literature describing their use and establishing or refuting their efficacy.

Sykes in 1986 performed a randomized, prospective, double-blinded study with 50 patients using topical nasal sprays with dexamethasone, tramazoline, and neomycin; dexamethasone and tramazoline without antimicrobial; and placebo. Both of the treatment groups showed improvement over placebo, but in those groups there was no significant difference in response rates between those patients receiving neomycin and those who did not. There were no adverse events reported. In the same year, Cuenant et al. reported success with neomycin-tixocortol irrigations in the treatment of chronic rhinosinusitis.

Scheinberg and Otsuji and Vaughn and Carvalho describe their use of various nebulized antimicrobials (including aminoglycosides) in patients with recurrent sinusitis. Both are uncontrolled, retrospective studies showing improvement in symptom scores. Neither study reported any major side effects. Leonard and Bolger describe a case report and review their success with the use of topical Ceftazidime in 50 patients. Only one patient reported stinging sensation during administration. They reported no problems with antibiotic resistance.

Studies by Davidson et al. , and Moss and King describe the use of topical antibiotics for sinusitis in patients with cystic fibrosis. They report improvement in sinusitis symptoms and reduction of need for revision sinus surgery in patients treated with surgery followed by topical intranasal tobramycin. They report no significant side effects.

Dudley described the use of topical gentamicin in a case report of a patient with atrophic rhinitis. The patient had resolution of her complaints without any adverse symptoms. He also describes a study by Thornell showing success with streptomycin nasal sprays and reports work by Rubinstein demonstrating safe administration of gentamicin into the nose without absorption by the nasal mucosa.

On balance, the literature describes topical antibiotics as a safe, but variably efficacious treatment for chronic rhinosinusitis. There is a paucity of prospective, randomized, blinded, and controlled studies. The purpose of this protocol is to describe a scientifically rigorous study of the use of broad spectrum antibiotic nasal sprays for chronic sinusitis.

The patient population for this study will consist of patients who have a history of multiple sinus infections each year that require treatment with antibiotics. The patients in this study will have had recurrent infections despite prior medical and surgical intervention. They will fulfill the criteria for chronic rhinosinusitis without nasal polyposis.

Treatment will include conventional treatment with oral antibiotics and a topical nasal steroid. In addition, patients will be randomized to receive either topical antibiotics or a vehicle placebo. The study will follow patients for a three month period.

Patients will be monitored for improvement in radiographic findings and quality of life when compared to a randomized and double-blinded placebo group. The patient population identified for inclusion in this study will also be evaluated for allergy and humoral and innate immunodeficiency. Nasal lavage will be obtained from the study population and pre and post-treatment comparisons will be performed.

DETAILED DESCRIPTION:
Chronic rhinosinusitis is a pervasive and costly disease. Recent estimates describe over 20 million Americans suffering from this diagnosis at a cost of over $4.3 billion per year. Primary intervention consists of oral antibiotics and nasal steroid sprays. A role for antifungal irrigation has also been proposed. Topical antibiotics are used by some physicians, but there are few reports in the published literature describing their use and establishing or refuting their efficacy.

Sykes in 1986 performed a randomized, prospective, double-blinded study with 50 patients using topical nasal sprays with dexamethasone, tramazoline, and neomycin; dexamethasone and tramazoline without antimicrobial; and placebo. Both of the treatment groups showed improvement over placebo, but in those groups there was no significant difference in response rates between those patients receiving neomycin and those who did not. There were no adverse events reported. In the same year, Cuenant et al. reported success with neomycin-tixocortol irrigations in the treatment of chronic rhinosinusitis.

Scheinberg and Otsuji and Vaughn and Carvalho describe their use of various nebulized antimicrobials (including aminoglycosides) in patients with recurrent sinusitis. Both are uncontrolled, retrospective studies showing improvement in symptom scores. Neither study reported any major side effects. Leonard and Bolger describe a case report and review their success with the use of topical Ceftazidime in 50 patients. Only one patient reported stinging sensation during administration. They reported no problems with antibiotic resistance.

Studies by Davidson et al. , and Moss and King describe the use of topical antibiotics for sinusitis in patients with cystic fibrosis. They report improvement in sinusitis symptoms and reduction of need for revision sinus surgery in patients treated with surgery followed by topical intranasal tobramycin. They report no significant side effects.

Dudley described the use of topical gentamicin in a case report of a patient with atrophic rhinitis. The patient had resolution of her complaints without any adverse symptoms. He also describes a study by Thornell showing success with streptomycin nasal sprays and reports work by Rubinstein demonstrating safe administration of gentamicin into the nose without absorption by the nasal mucosa.

On balance, the literature describes topical antibiotics as a safe, but variably efficacious treatment for chronic rhinosinusitis. There is a paucity of prospective, randomized, blinded, and controlled studies. The purpose of this protocol is to describe a scientifically rigorous study of the use of broad spectrum antibiotic nasal sprays for chronic sinusitis.

The patient population for this study will consist of patients who have a history of multiple sinus infections each year that require treatment with antibiotics. The patients in this study will have had recurrent infections despite prior medical and surgical intervention. They will fulfill the criteria for chronic rhinosinusitis without nasal polyposis.

Treatment will include conventional treatment with oral antibiotics and a topical nasal steroid. In addition, patients will be randomized to receive either topical antibiotics or a vehicle placebo. The study will follow patients for a three month period.

Patients will be monitored for improvement in radiographic findings and quality of life when compared to a randomized and double-blinded placebo group. The patient population identified for inclusion in this study will also be evaluated for allergy and humoral and innate immunodeficiency. Nasal lavage will be obtained from the study population and pre and post-treatment comparisons will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic rhinosinusitis symptoms present for greater than 12 weeks.
2. Two or more of the following symptoms:

   1. Anterior/posterior mucopurulent drainage
   2. Nasal obstruction
   3. Facial pain-pressure-fullness.
3. Endoscopy shows: within the past 3months prior to entry

   1. Discolored mucus or edema within the middle meatus or ethmoid region.
   2. Absence of polyps within the middle meatus.
4. Evidence of rhinosinusitis on CT scan within one year of study entry
5. History of prior sinus surgery with evidence of post-surgical changes on CT or clinical exam.
6. History of the following labs of: CH50, mannose binding lectin, quantitative immunoglobulin A, M, E and G, and titers for tetanus, diphtheria, and Streptococcus pneumoniae antibodies. If titers for tetanus, diphtheria, and Streptococcus pneumoniae are non-protective, then immunization will be performed and antibody titers will be reevaluated. If laboratory studies have not been done prior to entry the laboratory studies will be collected and performed during or post collection of study data to rule out any data from patients with known immunodeficiencies.
7. Skin prick testing will be performed at V1, unless done prior to study entry and is in the subjects medical record, for Dermatophagoides farinae, Dermatophagoides pteronyssinus, oak, bahia and bermuda grasses, cat, dog, ragweed, Alternaria, Aspergillus, American and German cockroach, and positive and negative controls.

Exclusion Criteria:

1. Allergy or adverse reaction to any of the medications intended for use in the study or any related compounds.
2. Receipt of systemic antibiotics for chronic rhinosinusitis within two weeks of beginning the study.
3. Receipt of systemic steroids within three months of beginning the study.
4. Patients using intranasal sympathomimetics or with evidence of rhinitis medicamentosa.
5. Sinus surgery within three months of starting study.
6. Smoking within one month of starting the study.
7. Pregnancy or lactation.
8. Primary ciliary dyskinesia, Sjogren's syndrome, Wegener's granulomatosis, atrophic rhinitis, cystic fibrosis, history of prior sinonasal malignancy, history of sinonasal irradiation, or other illness or treatment that might affect mucociliary transport within the nasal cavity or paranasal sinuses.
9. Clinically significant hepatic or renal disease.
10. Complicated sinusitis (e.g. Pott's puffy tumor, sinus malignancy, osteomyelitis, abscess, etc.)
11. Known immunodeficiency (including HIV, post transplant, diabetes).
12. Age less than 18 years of age.
13. Acute respiratory illness within 2 weeks of starting study.
14. Patients who meet the criteria for chronic rhinosinusitis with nasal polyps or allergic fungal rhinosinusitis.
15. Psychosocial issues that might preclude successful participation in the study.

V. Concomitant Medication/Treatment

In addition to use of the study drug or a vehicle-controlled placebo, the patient will be treated with Flonase 2 sprays each naris QD for the duration of the study. Rhinocort Aqua 4 sprays each naris QD will be substituted for patients with allergy or adverse reaction to Flonase. Augmentin 875mg PO BID will be given for 21 days beginning on the first day of the study period. Levaquin 500mg PO QD will be substituted for patients with allergy or adverse reaction to Augmentin. The patient will not use any adjunctive therapies such as oral or topical decongestants or antihistamines during the course of the study. No sinus or nasal surgery is planned during the course of the study. Patients who require additional treatment including surgery will be withdrawn from the study and considered treatment failures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
This is a prospective, randomized, double-blinded, placebo-controlled clinical study designed to evaluate the efficacy of topical antibiotics in treating chronic rhinosinusitis | 12 WEEKS

CONTACTS AND LOCATIONS:
Locations (1):
- USF, Tampa, Florida, United States